CLINICAL TRIAL: NCT00012012
Title: A Two Part Phase I/II Study Of Extended Field External Irradiation And Intracavitary Brachytherapy Combined With Chemotherapy And Amifostine In Carcinoma Of The Cervix With Positive Para-Aortic Or High Common Iliac Lymph Nodes
Brief Title: Radiation Therapy and Cisplatin With or Without Amifostine for Patients With Stage IIIB or IVA Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0116; CDR0000068472
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Cancer; Radiation Toxicity
Keywords: radiation toxicity; stage III cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries | interventions — Amifostine; ethanethiol; Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation therapy plus cisplatin (Experimental): Patients receive extended field external beam radiation therapy (RT) to the para-aortic region and pelvis, intracavitary brachytherapy with concurrent weekly cisplatin.
  Interventions: Drug: Cisplatin; Radiation: Intracavitary brachytherapy; Radiation: External beam radiation therapy
- Radiation therapy plus cisplatin and amifostine (Experimental): Patients receive extended field external beam radiation therapy (RT) to the para-aortic region and pelvis, intracavitary brachytherapy with concurrent weekly cisplatin and amifostine trihydrate.
  Interventions: Drug: Amifostine trihydrate; Drug: Cisplatin; Radiation: Intracavitary brachytherapy; Radiation: External beam radiation therapy

INTERVENTIONS:
Drug: Amifostine trihydrate — Amifostine will be delivered before each radiation treatment. Amifostine (500 mg) will be given as two equally-divided subcutaneous injections.
  Other Names: ethanethiol
  Arms: Radiation therapy plus cisplatin and amifostine
Drug: Cisplatin — Cisplatin will be given weekly with external beam radiation therapy and once with brachytherapy for a total of six doses. Patients receive 40 mg/m^2 by IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36.
Radiation: Intracavitary brachytherapy — For low dose rate (LDR) brachytherapy, cesium will be given in one to two intracavitary applications, within two weeks of completion of external radiation. The interval between the two applications will be one to three weeks. It is recommended that the total course of treatment be completed in less than eight weeks. High dose rate (HDR) brachytherapy may start as early as week two of external radiation. The minimum cumulative external and intracavitary dose should be 85 Gy.
Radiation: External beam radiation therapy — Patients will receive 1.8 Gy daily for five weeks for a total dose of 45 Gy; involved lateral parametrium and/or pelvic nodes should be boosted for a total dose (including intracavitary treatment) of 60 Gy ± 5%.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. Drugs such as amifostine may protect normal cells from the side effects of radiation therapy.

PURPOSE: Phase I/II trial to study the effectiveness of combining cisplatin and radiation therapy with or without amifostine in treating patients who have stage IIIB or stage IVA cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and tolerability of external beam radiotherapy, brachytherapy, and cisplatin in patients with para-aortic or high common iliac lymph node-positive carcinoma of the uterine cervix.
* Determine the feasibility and tolerability of this regimen with the addition of amifostine in these patients.
* Determine the efficacy of these 2 regimens, in terms of improving pelvic and para-aortic tumor control and distant metastases, in these patients.

OUTLINE:

* Phase I: Patients undergo external beam radiotherapy to the pelvis and para-aortic region 5 days a week for 5 weeks. Patients also undergo either intracavitary low-dose rate (LDR) brachytherapy in 2 applications beginning within 2 weeks after completion of external beam radiotherapy at 2-3 week intervals or 6 fractions of high-dose rate intracavitary brachytherapy over 8 weeks beginning as early as week 2 of external beam radiotherapy. Patients also receive cisplatin IV over 1 hour weekly for 6 weeks concurrently with external beam radiotherapy and once with LDR brachytherapy. Phase II proceeds only if toxicity in phase I is within expected parameters.
* Phase II: Patients receive external beam radiotherapy, brachytherapy, and cisplatin as in phase I. Patients also receive amifostine subcutaneously daily just before external beam radiotherapy and cisplatin. Treatment continues for up to 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven, locally advanced carcinoma of the uterine cervix

  * TNM classification stage IIIB or IVA
  * Disease metastatic to para-aortic or high common iliac lymph nodes

    * Prior complete surgical resection of involved lymph nodes or gross residual tumor involvement of a lymph node allowed
  * The following cellular types are eligible:

    * Squamous cell carcinoma
    * Adenocarcinoma
    * Adenosquamous carcinoma
  * The following cellular types are ineligible:

    * Small cell carcinoma
    * Carcinoid tumor
    * Glassy cell carcinoma
    * Clear cell carcinoma
    * Cystadenocarcinoma
* No metastatic disease outside of the pelvis (except to the para-aortic nodes)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* At least 6 months

Hematopoietic

* White blood cell count (WBC) at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* Alanine amino transferase (ALT) no greater than 2 times normal

Renal

* Creatinine no greater than 1.5 mg/dL (urinary diversion allowed)
* Corrected calcium normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent significant medical condition that would preclude study participation
* No insulin-dependent diabetes
* No other malignancy within the past 3 years except cutaneous basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic irradiation except transvaginal radiotherapy to control bleeding

Surgery

* See Disease Characteristics
* No prior tumor-directed surgery except lymph node biopsy/staging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-08; Primary Completion 2007-09 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Small, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (17):
- United States (17):
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Florida Oncology Associates at Southside Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Baptist Medical Center South, Jascksonville, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Akron City Hospital, Akron, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Viswanathan AN, Moughan J, Small W Jr, Levenback C, Iyer R, Hymes S, Dicker AP, Miller B, Erickson B, Gaffney DK. The quality of cervical cancer brachytherapy implantation and the impact on local recurrence and disease-free survival in radiation therapy oncology group prospective trials 0116 and 0128. Int J Gynecol Cancer. 2012 Jan;22(1):123-31. doi: 10.1097/IGC.0b013e31823ae3c9. PMID 22193645
- [Result] Small W Jr, Winter K, Levenback C, Iyer R, Hymes SR, Jhingran A, Gaffney D, Erickson B, Greven K. Extended-field irradiation and intracavitary brachytherapy combined with cisplatin and amifostine for cervical cancer with positive para-aortic or high common iliac lymph nodes: results of arm II of Radiation Therapy Oncology Group (RTOG) 0116. Int J Gynecol Cancer. 2011 Oct;21(7):1266-75. doi: 10.1097/IGC.0b013e31822c2769. PMID 21892091
- [Result] Small W Jr, Winter K, Levenback C, Iyer R, Gaffney D, Asbell S, Erickson B, Jhingran A, Greven K. Extended-field irradiation and intracavitary brachytherapy combined with cisplatin chemotherapy for cervical cancer with positive para-aortic or high common iliac lymph nodes: results of ARM 1 of RTOG 0116. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):1081-7. doi: 10.1016/j.ijrobp.2007.01.026. Epub 2007 Mar 29. PMID 17398031

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy Plus Cisplatin & Amifostine: Patients receive extended field external beam radiation therapy (RT) to the para-aortic region and pelvis, intracavitary brachytherapy with concurrent weekly cisplatin and amifostine trihydrate.
Period: Overall Study
Arm/Group | Radiation Therapy Plus Cisplatin | Radiation Therapy Plus Cisplatin & Amifostine
Started | 27 | 18
Completed | 26 | 15
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy Plus Cisplatin | Radiation Therapy Plus Cisplatin & Amifostine | Total
Number analyzed (Participants) | 26 | 15 | 41
Age, Continuous [Median (Full Range); unit: years] | 54 [30 to 76] | 56 [25 to 75] | 55 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 41
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Grade 3/4 Toxicity (Excluding Grade 3 Leukopenia)
Description: To determine the feasibility and tolerance of extended-field external radiotherapy to the pelvis and para-aortic region and intracavitary irradiation combined with weekly cisplatin using the rate of acute grade 3/4 toxicity rate (excluding grade 3 leukopenia). The first part of this study was designed to determine the acute grade 3/4 toxicity rate (excluding grade 3 leukopenia), to have a starting point for the second part (second arm) of the study.
Time Frame: From start of treatment to 90 days
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy Plus Cisplatin
Number analyzed (Participants) | 26
percentage of participants | 81 [66 to 96]

2. Primary Outcome: Number of Patients With Acute Grade 3/4 Toxicity (Excluding Grade 3 Leukopenia)
Description: The second part of this study (second arm) was designed to detect a 40% relative reduction (absolute from 77% to 46%) in the acute grade 3/4 toxicity (excluding grade 3 leukopenia) rate, with the addition of amifostine. A one-sided alpha of 0.05 and 80% power required 16 evaluable patients to detect the hypothesized difference. If ≤ 8 had the toxicity, it would be concluded that adding amifostine decreased this toxicity rate by at least 40%.
Time Frame: From start of treatment to 90 days
Population: All eligible patients
Measure: Number; unit: participants
Arm/Group | Radiation Therapy Plus Cisplatin and Amifostine
Number analyzed (Participants) | 15
participants | 13

3. Secondary Outcome: Pelvic Tumor Control
Time Frame: From registration to date of pelvic tumor failure or last follow-up. Analysis occurs after all patients have been potentially followed for 2 years.
Reporting Status: Not Posted

4. Secondary Outcome: Distant Metastases
Time Frame: From registration to date of distant mets or last follow-up. Analysis occurs after all patients have been potentially followed for 2 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE).
Arm/Group | Radiation Therapy Plus Cisplatin | Radiation Therapy Plus Cisplatin & Amifostine
Serious Adverse Events (participants affected / at risk) | 20/26 | 12/15
Other Adverse Events (participants affected / at risk) | 26/26 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Plus Cisplatin (N=26) | Radiation Therapy Plus Cisplatin & Amifostine (N=15)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 2 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 6 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Late RT Toxicity: Small/Lg Intestine: NOS (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 5 | 5
Vomiting NOS (Gastrointestinal disorders) | 5 | 4
Late RT Toxicity: Other: NOS (General disorders) | 2 | 1
Pain-other (General disorders) | 1 | 2
Infection NOS (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Leukopenia NOS (Investigations) | 2 | 3
Neutropenia (Investigations) | 2 | 1
Blood magnesium decreased (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 6 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis NOS (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Plus Cisplatin (N=26) | Radiation Therapy Plus Cisplatin & Amifostine (N=15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 | 15
Hearing-Other (Ear and labyrinth disorders) | 2 | 2
Abdominal pain NOS (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 8 | 5
Diarrhea NOS (Gastrointestinal disorders) | 15 | 14
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Late RT Toxicity: Small/Lg Intestine: NOS (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 13 | 10
Rectal bleeding (Gastrointestinal disorders) | 3 | 0
Vomiting NOS (Gastrointestinal disorders) | 7 | 8
Fatigue (General disorders) | 14 | 10
Late RT Toxicity: Other: NOS (General disorders) | 8 | 5
Pain due to radiation (General disorders) | 2 | 2
Pain-other (General disorders) | 6 | 3
Pyrexia (General disorders) | 2 | 3
Infection NOS (Infections and infestations) | 4 | 2
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 6 | 3
Late RT Toxicity: Skin (within the irradiated field): NOS (Injury, poisoning and procedural complications) | 4 | 2
Blood alkaline phosphatase NOS increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 5 | 5
Leukopenia NOS (Investigations) | 21 | 11
Lymphopenia (Investigations) | 3 | 3
Neutropenia (Investigations) | 12 | 8
Platelet count decreased (Investigations) | 17 | 9
Weight decreased (Investigations) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 7 | 3
Blood albumin decreased (Metabolism and nutrition disorders) | 4 | 4
Blood magnesium decreased (Metabolism and nutrition disorders) | 12 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 7 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 3
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 2
Late RT Toxicity: Bone: NOS (Musculoskeletal and connective tissue disorders) | 6 | 1
Dizziness (exc vertigo) (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 4
Dysuria (Renal and urinary disorders) | 6 | 1
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 8 | 3
Late RT Toxicity: Kidney: NOS (Renal and urinary disorders) | 5 | 2
Urinary frequency (Renal and urinary disorders) | 2 | 3
Pelvic pain NOS (Reproductive system and breast disorders) | 3 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 4
Menopausal symptoms (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.